CLINICAL TRIAL: NCT00101946
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of Nine-weeks Administration of Three Doses of SB-683699 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Nine-Weeks Treatment With 683699 In Subjects With Moderately-To-Severely Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683699/004
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Crohn's Disease
Keywords: CD; Crohn's Disease
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Drug: 683699

SUMMARY:
This study will evaluate the effectiveness and safety of the investigational drug 683699 in treating subjects with moderately to severely active CD (Crohn's Disease).

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with CD and reconfirmed in previous 2 years by a radiologic or endoscopic assessment including histology.
* CDAI (Crohn's Disease Activity Index) score of 220-450 after 1 week of screening.
* CRP (C-Reactive Protein) level of >4mg at screening.

Exclusion criteria:

* Significantly abnormal laboratory tests or ECG (electrocardiogram) results.
* Current use of an elemental diet or parenteral nutrition.
* Clinically significant positive stool culture.
* Ongoing neoplastic disease of the bowel.
* Bowel perforation other than fistulae.
* Has an ileostomy or colostomy.
* Fixed symptomatic gastrointestinal (GI) stricture within 6 months or obstructive symptoms within 3 months of screening.
* Any bowel resection within 12 months of screening or bowel resection without subsequent demonstration of recurrence of active CD.
* More than 100cm of bowel resected.
* Non-curative bowel surgery with 2 months of screening.
* Symptoms attributed to short bowel syndrome.
* Uncontrolled bacterial, viral, or fungal infection or congenital or acquired immunodeficiency.
* Women who are pregnant, breast feeding, or planning to become pregnant during the study.

Permitted medications:

* Less than or equal to 20mg/day oral corticosteroids for at least 4 weeks prior to screening and on stable doses for 2 weeks prior to screening.
* Azathioprine and 6-MP (6-Mercaptopurine) stable dose for 3 months prior to screening.
* 5-ASA (5-Aminosalicylic acid) stable dose for 1 month prior to screening.

Prohibited medications:

* Greater than 20mg/day oral corticosteroids, or systemic intravenous corticosteroids, or antibiotics as a treatment for CD within 4 weeks prior to screening.
* Cyclosporine or methotrexate during the 2 months prior to screening.
* Infliximab or other biological treatments within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who are responders at Week 6.

SECONDARY OUTCOMES:
- Proportion of subjects with response at other timepoints. - Proportion of subjects in remission. - Average rate of response for the CDAI score. - Mean change from baseline in CDAI score Improvement in Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (13):
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Houston, Texas
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan